CLINICAL TRIAL: NCT05254834
Title: The Vallania Study: A Case Control Study for the Development of Multiomics Blood Tests for Cancer Screening
Status: Completed | Type: Observational
Sponsor: Freenome Holdings Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: The Vallania Study/FRNM-008
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: Liquid Biopsy; Blood Test; Cancer Diagnostic; Genomics; Multiomics; Artificial Intelligence; Screening; Machine Learning; Freenome; Early Detection; Multicancer; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens will be de-identified and used to validate the performance characteristics of the Freenome test
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Cancer Group: Collect Subject Data Collect Blood Specimen
  Interventions: Diagnostic Test: Freenome Test
- Non-cancer Group: Collect Subject Data Collect Blood Specimen One Year Follow Up On Cancer Status
  Interventions: Diagnostic Test: Freenome Test

INTERVENTIONS:
Diagnostic Test: Freenome Test — Participants who provide informed consent, meet the eligibility criteria and provide a blood sample for this study will be enrolled.

SUMMARY:
This protocol is a case-control, multicenter, diagnostic study to collect blood samples to support the development of blood-based screening tests for multiple cancers.

ELIGIBILITY:
Key Inclusion Criteria:

* Age at least 30 years
* Able and willing to provide blood samples per protocol
* Able to comprehend and willing to sign and date the informed consent documents
* Participants must meet one of the following:

  * Diagnosed with a single primary cancer that has not yet been treated
  * No evidence or treatment of any cancer for at least 5 years prior to enrollment

Key Exclusion Criteria:

* A medical condition which, in the opinion of the investigator, should preclude enrollment in the study
* Known to be pregnant
* Any therapy for cancer, including surgery, chemotherapy, immunotherapy, and/or radiation therapy in the 5 years preceding enrollment
* Participated or currently participating in a clinical research study in which an experimental medication has been administered in the last 30 days
* Participated in or currently participating in another Freenome clinical study
* For the control cohort: Any previous cancer diagnosis in the 5 years preceding enrollment, or recurrence of the same primary cancer within any timeframe; or concurrent diagnosis of multiple primary cancers within any timeframe
* For the cancer cohorts: Any previous cancer diagnosis in the 5 years preceding enrollment, apart from the current cancer diagnosis; OR recurrence of the same primary cancer within any timeframe; OR concurrent diagnosis of multiple primary cancers within any timeframe

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 30+ who have been newly diagnosed (treatment-naive) with cancer and Adults 30+ without cancer
Sampling Method: Non-Probability Sample
Enrollment: 7435 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Comparison of Blood Samples from Cancer Case and Non-cancer Control Participants | 12 months
  To compare blood samples from cancer case and non-cancer control subjects in order to develop and characterize blood-based multiomics tests in specific cancer types or in a combination of multiple cancers.

CONTACTS AND LOCATIONS:
Locations (68):
- United States (68):
  - Central Alabama Research, Birmingham, Alabama
  - Alabama Oncology, Birmingham, Alabama
  - Honor Health, Scottsdale, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - John Muir Health, Concord, California
  - Carbon Health, Corona, California
  - Miller Bioconnect, El Cajon, California
  - Gastroenterology and Liver Institute, Escondido, California
  - Women's Cancer Network, Fresno, California
  - San Diego Clinical Trials, La Mesa, California
  - Urology Alliance Clinical Research, Los Angeles, California
  - Mercy Cancer Center, Merced, California
  - Pomona Valley Hospital Medical Center/Cancer Care Center, Pomona, California
  - St. Mary's Medical Center, San Francisco, California
  - Dominican Hospital Dignity Health, Santa Cruz, California
  - Stockton Hematology Oncology, Stockton, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Eastern CT Hematology and Oncology Associates, Norwich, Connecticut
  - RecioMed Clinical Research, Boynton Beach, Florida
  - Mid Florida Hematology & Oncology Center, Orange City, Florida
  - Emerald Coast OBGYN, Panama City, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Cancer Center of Middle Georgia (QCCA), Dublin, Georgia
  - Specicare, Gainesville, Georgia
  - University of Chicago, Chicago, Illinois
  - Northwest Oncology & Hematology, Rolling Meadows, Illinois
  - Objective Health Network (Digestive Research Alliance of Michiana, LLC), South Bend, Indiana
  - Ascension Via Christi Hospital, Wichita, Wichita, Kansas
  - Saint Joseph Cancer Center, Lexington, Kentucky
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Ascension Providence Rochester Hospital, Rochester Hills, Michigan
  - Covenant HealthCare, Saginaw, Michigan
  - University of Minnesota, School of Public Health, Environmental Health Sciences, Minneapolis, Minnesota
  - Central Care Cancer Center, Bolivar, Missouri
  - Billings Clinic, Billings, Montana
  - Logan Health Research, Kalispell, Montana
  - Cancer Care Specialists Reno, Reno, Nevada
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - NYU, New York, New York
  - NY Cancer & Blood Specialists, Port Jefferson Station, New York
  - White Plains Hospital, White Plains, New York
  - Altru Health System, Grand Forks, North Dakota
  - Gabrail Cancer Center Research, Canton, Ohio
  - Objective Health Network, Dayton, Ohio
  - Hightower Clinical Research, Oklahoma City, Oklahoma
  - St. Charles Health System, Inc, Bend, Oregon
  - Doylestown Health, Doylestown, Pennsylvania
  - Pennsylvania Cancer Specialists & Research Institute, Gettysburg, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Donald Guthrie Foundation, Sayre, Pennsylvania
  - USDH Clinical Research, Wyomissing, Pennsylvania
  - Cancer Care Associates of York (QCCA), York, Pennsylvania
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - ObjectiveHealth, Inc, Franklin, Tennessee
  - Christus Spohn Shoreline Hospital, Corpus Christi, Texas
  - Oncology Consultants, Houston, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
  - Centra Lynchburg Hematology Oncology, Lynchburg, Virginia
  - Objective Health Network, Richmond, Virginia
  - Northwest Medical Specialties (QCCA), Tacoma, Washington
  - SSM Health-Dean Medical Group, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No